CLINICAL TRIAL: NCT06717139
Title: Recurrence and Predictive OCT Biomarkers in Neovascular Age Related Macular Degeneration After Discontinuation of Anti-VEGF Therapy
Brief Title: Recurrence and Predictive OCT Biomarkers in Quiescent Neovascular AMD
Status: Active, not recruiting | Type: Observational
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Anders Kvanta, MD, PhD, professor, St. Erik Eye Hospital
Other Study IDs: StErik
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Retinal Diseases; Macular Degeneration; Neovascular (Wet) Age-Related Macular Degeneration
Keywords: AMD; biomarker; recurrence; OCT
MeSH Terms: conditions — Retinal Diseases; Macular Degeneration; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Age-related macular degeneration (AMD) is the most common cause of severe visual impairment and blindness in elderly patients. The central part of the retina is called the macula and is very important for visual acuity. In wet AMD, blood vessels grow under the macula and leak fluid, which leads to swelling in the macula and vision loss. Patients who develop wet AMD are treated with injections into the eye. Today, the treatment can be stopped when the patient has reached an interval of six months between the injections, without showing any signs of disease activity. However, it is not unusual for the swelling in the macula to return and the injections then must be resumed. Today, it is not known exactly how many patients suffer from active disease recurrence, or at what point of time the recurrence usually happens. Furthermore, it remains unclear which patients are at a higher risk of active disease recurrence.

Optical coherence tomography (OCT) is a simple and quick measurement method, similar to taking a photograph of the inside of the eye, to investigate whether there is swelling or other changes in the macula. With OCT, the retina is measured with infrared light. With OCT angiography (OCT-A), which is done in the same simple way, it is also possible to visualize the diseased blood vessels and other changes in the retina.

Under the retina is the choroid layer of the eye, OCT can also be used to measure the thickness and circulation of the choroid.

No large prospective studies have investigated changes on OCT, changes in the diseased vessels on OCT-A, choroidal thickness and choroidal circulation on OCT, and the risk of recurrence of disease requiring treatment in wet AMD.

The study will be conducted as a prospective study at St. Erik's Eye Hospital, a total of 220 patients with wet AMD, where the treatment interval has been extended to 6 months without signs of disease activity, will be included in the study and followed for 18 months, i.e. up to two years after the last injection. Patients with disease recurrence during the follow-up period will be withdrawn from the study and resume treatment.

The aim of the study is to see if there is a relationship between specific changes on OCT and OCT angiography and later recurrence in wet AMD, to investigate how many patients experience disease recurrence and to find out when the recurrence usually occurs. No previous prospective study has investigated these different parameters.

Increased knowledge of how many patients experience recurrence of wet AMD requiring treatment, as well as a deeper understanding of which patients are at greater risk of recurrence, could have a major impact on the planned follow-up in this population. Furthermore, by improving the conditions for being able to identify recurrences earlier, the risk of irreversible vision loss could also decrease in this patient group.

DETAILED DESCRIPTION:
Biomarkers predicting recurrence risk in patients with quiescent neovascular AMD

Background Age-related macular degeneration (AMD) is the leading cause of visual impairment and blindness among older individuals. There are two types of AMD. Dry macular degeneration is the most common type and usually progress slowly over time. Dry AMD can progress to wet (neovascular) macular degeneration, which is characterized by blood vessels that grow under the retina and leak fluid. The wet type is more likely to cause a relatively sudden change in vision resulting in serious vision loss.

The diagnostic procedure in neovascular AMD involves an assessment of the macular edema and other structural changes of the macula with Optical Coherence Tomography (OCT), which is a measurement with infrared light of the different layers of the retina. Previously the standard procedure to diagnose wet AMD was performing an angiography with administration of intravenous fluorescein. Today it is possible to visualize the neovascular vessels in wet AMD with OCT-angiography (OCT-A) which is non-invasive and also considerably faster to perform.

With the introduction of intravitreal anti-VEGF-injections 20 years ago, the visual outcome for AMD patients has improved substantially. After a loading dose of anti-VEGF the patient is generally followed and treated according to a treat-and-extend regimen, until the macula remains dry for a longer interval and treatment may be discontinued.

During the last decade the frequency of anti-VEGF injections has grown exponentially, now causing a considerable economic burden and a great logistic challenge for the ophthalmological community and the health care services. , It is therefore of great interest to investigate the discontinuation of therapy in patients that have shown disease stability over extended periods. A recent prospective study showed that 53% of the patients had recurrent macular edema during the first year after treatment was discontinued. However, only 41% of these patients experienced symptoms of visual loss or metamorphopsia at the time of recurrence. This study also showed that patients with a pigment epithelium detachment (PED) had a 74% recurrence rate compared with 48% in patients without a PED, during the first year after treatment discontinuation. It is of great interest predicting which patients are at higher risk of disease recurrence.

Previous studies have shown that the localization of the fluid in wet AMD is relevant for the visual prognosis. Intraretinal fluid is strongly associated with active disease and has a negative impact on visual prognosis. Subretinal fluid on the other hand, may not have a significant negative effect on visual acuity, and is associated with better anatomical and functional outcome with a lower risk of progression towards geographic atrophy than intraretinal fluid. Subretinal fluid may be a sign of RPE dysfunction alone and is not necessarily a sign of active disease or neovascular AMD, therefore some degree of subretinal fluid that has been categorized as refractory, is generally accepted in the treatment of wet AMD.

After treatment with anti-VEGF agents both the lesion area and the vessel density decrease significantly on OCT-A. However, the caliber of the main feeder vessel seems more resistant to treatment and may not be affected. Larger feeder vessels may be more resistant to anti-VEGF therapy due to the presence of overlying pericytes that do not surround the smaller vessel branches of the vascular membrane.

OCT can also be used to assess the choroidal perfusion by measuring the choroidal thickness (CT) and the choroidal vascularity index (CVI), which is a tool for assessing the vascular network with enhanced depth imaging OCT. Some studies suggest that inadequate choroidal perfusion may lead to hypoxia of the retinal pigment epithelium (RPE) and increased VEGF production and the formation of neovascular vessels, hence increasing the risk for disease activity. There may also be a correlation between an increase in CT and disease recurrence of neovascular AMD, suggesting that CT could potentially be used as a monitoring tool in AMD management.

No larger prospective studies have investigated the characteristics of the lesion structure on OCT-A and the choroidal perfusion on OCT, and the risk of disease recurrence in wet AMD.

Purpose and aims

Primary endpoint:

• To investigate the impact of the following OCT-A and OCT biomarkers on the risk of disease recurrence in wet AMD:

* Neovascular lesion area, largest lesion diameter, largest vessel diameter, presence of anastomosis and loop patterns and vessel density on OCT-A
* CT and CVI on EDI-OCT
* The presence of a PED and PED size on OCT

Secondary endpoints:

* To assess the time to recurrence and the number of patients with recurrence during a 2-year period after discontinued treatment.
* To investigate if there is a correlation between disease recurrence and the total number of given injections, time elapsed since start of treatment, previous episodes of recurrence, age, gender, MNV type (MNV type 1, 2, 3 or PCV) and the presence of vitreomacular traction or adhesion, geographic atrophy and submacular fibrosis.
* To investigate if minor subretinal edema (≤50 µm), that has been classified as non-active disease, at baseline is a risk factor for disease recurrence.
* To assess the change in foveal thickness (CST) on OCT over time.
* To assess the change in visual acuity measured in ETDRS over time.

Hypothesis In neovascular AMD, choroidal perfusion on OCT and lesion characteristics on OCT-A may correlate with the risk of disease recurrence after discontinued treatment with anti-VEGF. The presence of a PED at the time of treatment discontinuation is a risk factor for disease recurrence.

Project description The study will be carried out as a prospective study at St. Erik Eye Hospital at the department of vitreoretinal diseases. A total of 220 patients will be included in the study and followed for 18 months.

Inclusion criteria: Patients with wet AMD previously followed and treated according to a "treat and extend" regimen, reaching intervals of 24-32 weeks without any evidence of disease activity on OCT, and BCVA ≥35 letters (Snellen 20/200) and near vision at least 24 points and age 55 years or older are eligible for study inclusion.

Exclusion criteria: wet AMD with signs of disease activity (neovascular exudative intraretinal fluid or significant subretinal fluid on OCT, or macular bleeding or exudation on fundus exam). Other coexisting causes for macular edema than AMD (for example central serous chorioretinopathy, retinal vein occlusion or diabetic macular edema).

Patients that are eligible for study inclusion will be examined at baseline 6 months (24-32 weeks) after the last treatment with anti-VEGF, and then monitored for disease recurrence quarterly for 18 months (month 3, 6, 9, 12, 15, 18), meaning that the final study visit will take place 24 months after the last anti-VEGF injection.

Best corrected visual acuity (measured in ETDRS) and near vision will be tested at each study visit. A complete slit lamp ophthalmic examination will be performed at each study visit after administration of dilating eye drops.

OCT will be performed at each study visit to evaluate any signs of recurrence and to assess morphological changes in the macula (including PED and VMT/VMA). EDI-OCT will be performed at baseline and at the end of study to measure the CT and to assess the CVI. An automated OCT software will be used to assess the CVI.

OCT-A will be performed at each study visit to measure the lesion area and diameter and the lesion vessel diameter, other morphological changes of the neovascular lesion will also be assessed. If there is no visible neovascular membrane on OCT-A at baseline this will also be documented.

Angiographic subtype of the neovascular membrane (type 1 MNV, type 2 MNV, type 3 MNV or polypoidal choroidal vasculopathy) will also be determined based on OCT-A at baseline, and if necessary on previous OCT-A performed at diagnosis, and/or previously performed retinal angiography (fluorescein and indocyanine green).

In case of disease recurrence (relapsing macular edema on OCT and/or findings corresponding to macular bleeding or exudates) the patient will be excluded from the study protocol and treated and followed according to current guidelines. However, a study visit will take place at the time of the planned final study visit, 18 months after baseline, in these patients.

Statistical analysis The relationship between the risk of relapse in wet AMD and the presence of almost all the biomarkers investigated in the study has not been previously established. It is therefore not possible to estimate a general sample size based on previous study results. A previous study showed that patients with PED at baseline had a 74% risk of relapse compared to 48% in patients without PED. Assuming, based on these results, a proportional recurrence rate of 70% versus 50% with and without a particular biomarker, respectively, with a statistical power of 80% and a p value of <0.05, a population of 93 patients would be required. Assuming a dropout rate of at least 10%, 105 patients need to be included in the study. However, because of the lack of previous study data on biomarkers and the risk on recurrence, and to ensure statistically significant results, the investigators will include 220 patients in the study. Based on previous patient flow data at St. Erik Eye Hospital, inclusion will take approximately 18 months.

Data analysis will be performed with the SPSS statistical software. For statistical data analysis, the independent Student's t-test will be used for continuous variables and the Chi-Square test / Fisher's Exact Test will be used for categorical data. For continuous variables mean ± SD will be used and counts with percentages for categorical variables. A P-value less than 0.05 will be considered statistically significant. A multivariate regression analysis will be used to evaluate the association between the baseline biomarkers and the risk for recurrent disease adjusting for potential confounders.

Ethical considerations No treatment will be given in the study. This is an observational prospective study, the study participants will be followed more frequently and for a longer period of time, compared to standard procedure. The investigators will therefore have the possibility to detect any sign of disease recurrence earlier than otherwise, and the patient will then be offered treatment according to current guidelines. All patients with wet AMD without disease activity or other causes for macular edema at baseline will be offered to participate in the study. If disease activity can be identified at baseline the patient will receive continued treatment and follow up according to current guidelines.

Significance OCT and OCT-A are non-invasive examinations that are quick and easy to perform and can provide information on biomarkers that may serve as monitoring and predictive tools for disease recurrence in neovascular AMD. A deeper understanding of which patients have a higher risk of recurrence could have a significant impact on the follow-up schedule in patients that have previously shown disease stability over extended periods of time. Identifying these patients would be of great value considering the great economic burden and growing logistic challenge in AMD patient care.

By establishing relevant biomarkers and thereby providing easily accessible tools to identify which patients have a higher risk of recurrence, this patient group can be followed more frequently after discontinued treatment, also making it possible to identify possible recurrence and resume treatment earlier in these patients, which may have a positive effect on the visual prognosis, by avoiding delayed diagnosis and possible non-reversible vision loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with wet AMD previously followed and treated according to a "treat and extend" regimen, reaching intervals of 24-32 weeks without any evidence of disease activity on OCT, and BCVA ≥35 letters (Snellen 20/200) and near vision at least 24 points and age 55 years or older are eligible for study inclusion.

Exclusion Criteria:

* wet AMD with signs of disease activity (neovascular exudative intraretinal fluid or significant subretinal fluid on OCT, or macular bleeding or exudation on fundus exam). Other coexisting causes for macular edema than AMD (for example central serous chorioretinopathy, retinal vein occlusion or diabetic macular edema).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 220 patients that have been treated with intraviteral anti-VEGF injections for neovascular AMD at the retinal clinic at St Erik Eye Hospital, Stockholm, Sweden.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2026-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
The association between OCT and OCTA biomarkers and disease recurrence in neovascular AMD | From enrollment to the end of study at 18 months
  To investigate the impact of the following OCT-A and OCT biomarkers on the risk of disease recurrence in wet AMD:
  * Neovascular lesion area, largest lesion diameter, largest vessel diameter, presence of anastomosis and loop patterns and vessel density on OCT-A
  * CT and CVI on EDI-OCT
  * The presence of a PED and PED size on OCT

CONTACTS AND LOCATIONS:
Locations (1):
- St Erik Eye Hospital, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
A decision has not yet been made